CLINICAL TRIAL: NCT03952442
Title: The Effect of Nutrition Education Program on the Nutrition Status and Life Quality of Postoperative Patients With Gastric Cancer
Brief Title: Nutrition Education Program for Postoperative Patients With Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-211
Record Dates: First submitted 2019-05-05; First posted 2019-05-16 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Gastric Cancer; Nutrition Disorders
Keywords: gastric cancer; nutrition; health education
MeSH Terms: conditions — Stomach Neoplasms; Nutrition Disorders; Health Education

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: routine nutrition education
- experimental group (Experimental)
  Interventions: Other: standardized nutrition education

INTERVENTIONS:
Other: standardized nutrition education — Give nutrition health education every two weeks and regular survey and intervention. The education booklets are made based on the guideline and characteristics of the disease.
  Arms: experimental group
Other: routine nutrition education — Give nutrition education if the patient visits the clinics. Irregular survey and intervention were given to the patients.
  Arms: control group

SUMMARY:
Using randomized control study, explore the effect of standardized nutrition education program on the nutrition status and life quality of patients with gastric cancer after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with gastric cancer and receive operation.
* Patients need nutrition support treatment
* Informed consent.

Exclusion Criteria:

* Critical patients or stage IV
* Patients with severe hepatic cirrhosis, Chronic Obstructive Pulmonary Disease, chronic renal failure, intestinal obstruction, stroke.
* Unconscious or psychiatric patients
* Patients with communication problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
risk of malnutrition | Week 0
  Nutrition Rsik Screening 2002 is used to assess the risk of malnutrition.
risk of malnutrition | Week 12
  Nutrition Rsik Screening 2002 is used to assess the risk of malnutrition.
BMI | Week 0
  Body mass index is a measure of body fat based on height and weight that applies to adult men and women. It equals to weight divided by height square.
BMI | Week 12
  Body mass index is a measure of body fat based on height and weight that applies to adult men and women. It equals to weight divided by height square.
albumin | Week 0
  level of serum albumin
albumin | Week 12
  level of serum albumin
Quality of Life (QOL) | Week 0
  The QOL was measured by the European Organization for Research and Treatment quality of life version 3 questionnaire (EORTC QLQ-C30) simplified Chinese version. It contains five functional scales (physical, role, cognitive, emotional, and social), three symptoms scales (fatigue, pain, and nausea and vomiting), a global health scale, a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, appetite loss, insomnia, constipation, and diarrhea) and financial impact of the disease. For most items, four response categories from 1 (not at all) to 4 (very much) are employed; two items (overall health, overall quality of life) have response categories ranging from 1 to 7. A high scale score represents a higher response level. Thus a high score for a functional scale, the global health status or overall QOL represents a high or healthy status or a high QOL; however, a high score for the symptom scales represents a high level of symptom.
Quality of Life (QOL) | Week 12
  The QOL was measured by the European Organization for Research and Treatment quality of life version 3 questionnaire (EORTC QLQ-C30) simplified Chinese version. It contains five functional scales (physical, role, cognitive, emotional, and social), three symptoms scales (fatigue, pain, and nausea and vomiting), a global health scale, a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnea, appetite loss, insomnia, constipation, and diarrhea) and financial impact of the disease. For most items, four response categories from 1 (not at all) to 4 (very much) are employed; two items (overall health, overall quality of life) have response categories ranging from 1 to 7. A high scale score represents a higher response level. Thus a high score for a functional scale, the global health status or overall QOL represents a high or healthy status or a high QOL; however, a high score for the symptom scales represents a high level of symptom.

SECONDARY OUTCOMES:
physical function status | Week 0
  Using Eastern Cooperative Oncology Group to assess the physical function.
physical function status | Week 12
  Using Eastern Cooperative Oncology Group to assess the physical function.
Knowledge-Attitude-Practice | Week 12
  Knowledge Scale composes of 10 questions and 10 scores for each question. Attitude and Practice Scale have 5 questions. Each question is rated as A、B、C. A represents 20 score and B is 10 score.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No